CLINICAL TRIAL: NCT01902238
Title: EUS-guided Ethanol-lipiodol Ablation of Pancreatic Neuroendocrine Tumor: a Prospective Feasibility and Long Term Outcome
Brief Title: EUS-guided Ethanol-lipiodol Ablation of Pancreatic Neuroendocrine Tumor: a Prospective Study
Acronym: EUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Dankook University (Other)
Responsible Party: Principal Investigator, Do Hyun Park, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NET ETHANOL
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Efficacy; Safety; Feasibility
Keywords: neuroendocrine tumor; ethanol; endoscopic ultrasonography
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-guided ethanol-lipiodol mixture ablation (Experimental): By using 3D-volumetric analysis, the optimal volume of ethanol is calculated by computer estimation of areas on each axial image, using EUS software permitting volume calculation. After calculating optimal ethanol volume by 3D volumetric analysis, we advance the needle into the tumor and inject estimated volume of ethanol/lipiodol (1:1 mixture), typically 1 to 1.5 ml.
  Interventions: Procedure: EUS-guided ethanol-lipiodol mixture ablation

INTERVENTIONS:
Procedure: EUS-guided ethanol-lipiodol mixture ablation — By using 3D-volumetric analysis, the optimal volume of ethanol/lipiodol (1:1 mixture) is calculated by computer estimation of areas on each axial image, using EUS software permitting volume calculation. After calculating optimal ethanol volume by 3D volumetric analysis, we advance the needle into the tumor and inject estimated volume of ethanol, typically 1 to 1.5 ml.

SUMMARY:
The present study evaluate the safety and efficacy of EUS-guided ethanol-lipiodol ablation for the treatment of pancreatic NET

DETAILED DESCRIPTION:
Pancreatic neuroendocrine tumor, including insulinoma, increasingly are being encountered in clinical practice. Management of pancreatic NET is challenging because most are asymptomatic but may have malignant potential, and surgical resection of pancreatic neoplasm is associated with substantial morbidity of 20%-40% and a mortality rate of 2%. Management strategy needs to be individualized, applying a risk-benefit analysis to each patient. Recently, pancreatic tissue ablation by EUS-guided injection of ethanol or other chemotherapeutic agents can be performed safely, with few procedure-related complications. Levy et al. demonstrated that EUS-guided ethanol ablation for insulinoma was both safe and feasible, and symptomatic improvement was achieved in 8 of 8 patients (100%). However, previous study have included only a small number of patients and evaluated only short-term outcomes. In addition, lipiodol permits the drug to concentrate in the tumor. To obtain an embolic effect and prevent washout of the ethanol, ethanol/lipiodol mixture is administered into the tumor. The present study evaluate the safety and efficacy of EUS-guided ethanol-lipiodol ablation for the treatment of pancreatic NET

ELIGIBILITY:
Inclusion Criteria:

* Pancreas NET(including insulinoma) < 2cm in diameter
* Poor surgical candidate (involving the head of the pancreas or multifocal NET, advanced comorbidity, age >75 years of age)
* Refuse to surgery

Exclusion Criteria:

* Younger than 18 years of age
* Coagulopathy (INR >1.5, Platelet <50,000)
* Evidence of active pancreatitis
* Inability to safely undergo EUS
* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment response | more than 3 years after procedure
  Final tumor viability will be assessed using contrast enhanced CT, and EUS-guided FNA at 3 years after procedure

SECONDARY OUTCOMES:
The number of participants with post-procedure adverse events | until 3 months after procedure
  Adverse events were defined as any procedure-related complications during the procedure or within 3 months, including pancreatitis, bleeding, and peripancreatic fluid collection

OTHER OUTCOMES:
Technical feasibility | at the time of procedure
  Technical success was defined as the ability to access and inject the mixture of ethanol/lipiodol into target tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Study Director — Asan Medical Center, Seoul, Korea, Republic of
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No